CLINICAL TRIAL: NCT00002062
Title: Open-Label "Compassionate" Use Study of Spiramycin for the Treatment of Diarrhea Due to Chronic Cryptosporidiosis in Immunocompromised Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhone-Poulenc Rorer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 011A; CCA 901
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-10

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Spiramycin; AIDS-Related Opportunistic Infections; Immune Tolerance; Cryptosporidiosis; Diarrhea; Drugs, Investigational; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; AIDS-Related Opportunistic Infections; Diarrhea; Acquired Immunodeficiency Syndrome | interventions — Spiramycin

INTERVENTIONS:
Drug: Spiramycin

SUMMARY:
This protocol provides for the availability of spiramycin under compassionate-use conditions for the treatment of chronic diarrhea due to cryptosporidium in patients with a compromised immune system, thus deriving additional information regarding its safety and efficacy profile.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with known sensitivity to macrolide antibiotics are excluded. Consideration must be given to the fact that spiramycin is a macrolide antibiotic and, therefore, may have the potential to induce hepatotoxicity.

* Patients with a compromised immune system may have hepatic abnormalities or even hepatitis. If the benefit-to-risk ratio does not favor the use of spiramycin, the patients must be excluded from the study.

Concurrent Medication:

Excluded:

* Other investigational drugs.

Patients with known sensitivity to macrolide antibiotics are excluded. Consideration must be given to the fact that spiramycin is a macrolide antibiotic and, therefore, may have the potential to induce hepatotoxicity.

* Patients with a compromised immune system may have hepatic abnormalities or even hepatitis. If the benefit-to-risk ratio does not favor the use of spiramycin, the patients must be excluded from the study.

Prior Medication:

Excluded within 7 days of study entry:

* Other investigational drugs.

Diagnosis of chronic diarrhea due to cryptosporidiosis and a compromised immune system but not limited to patients with AIDS.

* Patients receiving chemotherapy for a malignancy.
* Patients who are iatrogenically immune-suppressed following organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Rhone - Poulenc Rorer Pharmaceuticals, Horsham, Pennsylvania, United States